CLINICAL TRIAL: NCT05540015
Title: Use of Erbium Laser With the Wavelength 2.94 nm for Extraction of the Impacted Lower Third Molars
Brief Title: Use of Erbium Laser for Extraction of the Third Molars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6482963527
Record Dates: First submitted 2022-09-09; First posted 2022-09-14 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Third Molar Extraction; Impacted Third Molar Tooth
Keywords: Impacted third molars; Erbium laser; Atraumatic extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group with impacted third molar, extracted by cutting and rotary tools (Active Comparator): The study group will include 28 patients with indications (impacted third molars that exerts pressure on the adjacent tooth and cause inflammation process in the surrounding tissue; absence of antagonist; pericorinitis; periodontitis; periodontal pockets) for the impacted third molar extraction. Patients will be comparable by gender and age, the patients age will be between 18 and 70 years. Patients should be with therapeutic and surgical oral hygiene and without co-morbidities.
  Interventions: Procedure: Third molar extraction by cutting and rotary tools
- Group with impacted third molar, extracted by erbium laser 2.94 nm (Active Comparator): The study group will include 28 patients with indications (impacted third molars that exerts pressure on the adjacent tooth and cause inflammation process in the surrounding tissue; absence of antagonist; pericorinitis; periodontitis; periodontal pockets) for the impacted third molar extraction.Patients will be comparable by gender and age, the patients age will be between 18 and 70 years. Patients should be with therapeutic and surgical oral hygiene and without co-morbidities.
  Interventions: Procedure: Third molar extraction by erbium laser with wavelength 2.94 nm

INTERVENTIONS:
Procedure: Third molar extraction by cutting and rotary tools — Extraction of the impacted lower third molar will be conducted using cutting and rotary tools under the local anesthesia (Ultracain D-S 1:100000 40 mg/ml, active substance- articaine+epinephrine, registration № П N015119/01 ). Scalpel will be used for the incision of the soft tissues, rotary instruments will be used for the bone tissue and tooth fragmentation. After the extraction the wound will be sutured by the suture material.
  Arms: Group with impacted third molar, extracted by cutting and rotary tools
Procedure: Third molar extraction by erbium laser with wavelength 2.94 nm — Extraction of the impacted lower third molar will be conducted using erbium laser with wavelength 2.94 nm under the local anesthesia (Ultracain D-S 1:100000 40 mg/ml, active substance- articaine+epinephrine, registration № П N015119/01 ). The soft tissue and bone tissue will be dissected by erbium laser with wavelength 2.94 µm (Erbium laser Smart 2940D plus with the wavelength 2,94 µm, company- DEKA, Italy, registration № 2005/1245). After the extraction the wound will be sutured by the suture material (registration № ФСЗ 2010/06040; 07.08.2018)
  Arms: Group with impacted third molar, extracted by erbium laser 2.94 nm

SUMMARY:
A comparative analysis of the effectiveness of the erbium laser with the wavelength of 2.94 µm and traditional instruments in the extraction of the impacted lower third molars will be performed. Clinical, radiological and biochemical findings will be assessed after extraction of the impacted lower third molars.

DETAILED DESCRIPTION:
A single-centre, interventional, non-randomized, prospective clinical trial in 2 parallel groups is planned. The lower third molars will be extracted in 60 patients. There will be 2 groups. The number of men and women in both groups will be the same, the patients age will be between 18 and 70 years. In the study group the lower third molars will be extracted using erbium laser with a wavelength of 2.94 µm (Erbium laser Smart 2940D plus with the wavelength 2,94 µm, company- DEKA, Italy, registration № 2005/1245), in the control group the lower third molars will be extracted using the conventional method (cutting and rotating instruments). Postoperative clinical symptoms such as collateral soft tissue swelling, postoperative pain, trismus in the extraction site and healing time (epithelization and bone regeneration) will be assessed. The epithelization will be assessed after 7, 10, 14 days. The bone regeneration will be assessed by cone beam computed tomography (KAVO, ORTHOPANTOMOGRAPH ОР 3D, type: РСХ-1; registration № РЗН 2020/10586) after 1, 3, 6 months. The radiation exposure will not exceed the permissible limits. Biochemical indicators in the saliva will be assessed before extraction, after extraction, 3 days and 7 days after the extraction. The Shapiro-Wilk test will be applied to check the normality of variable distribu- tion. Qualitative variables will be analyzed by Pearson's chi-squared test. Quantitative variables (normal distribution of variable) will be analyzed by Students t-test, non-normal distribution of variables will be analyzed by Mann-Whitney U test.

ELIGIBILITY:
Inclusion Criteria:

1. Signing of written informed consent of the patient to participate in a study
2. Age from 25 to 50 years old
3. Indications for impacted third molar extraction
4. Patients who are medically stable
5. Therapeutic and surgical oral hygiene before surgery (absence of inflammatory diseases, caries, pulpitis, periodontitis in oral cavity)

Exclusion Criteria:

1. Refusal of the patient from further participation in the study
2. Pregnancy diagnosed after the inclusion into the trial
3. Non-compliance by the patient with postoperative recommendations
4. Absence of a lower second molar

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Assessment the level of bone regeneration according to Radiographic bone height (RBH) | Days 180 after extraction
  Assessment the level of bone regeneration according to Radiographic bone height (RBH) by cone beam computed tomography after extraction of the lower third molar. (Radiographic bone height (RBH)- is the distance between root apex of the distal root and uppermost intersecting point between distal root of the second molar and mesial wall of extraction socket, it will be measured on the cone beam computed tomography)

SECONDARY OUTCOMES:
Radiographic bone height (RBH) | 3;6 months
  Assessment the level of bone regeneration according to Radiographic bone height (RBH) by cone beam computed tomography after extraction of the lower third molar with erbium laser. (Radiographic bone height (RBH)- is the distance between root apex of the distal root of the second molar and uppermost intersecting point between distal root of the second molar and mesial wall of extraction socket, it will be measured on the cone beam computed tomography)
Radiographic infrabony defect (RID) | 3;6 months
  Assessment the level of bone regeneration according to Radiographic infrabony defect (RID) by cone beam computed tomography after extraction of the lower third molar with erbium laser. (Radiographic infrabony defect (RID) is the distance between cemento-enamel junction of the second molar and uppermost intersecting point between distal root of the second molar and mesial wall of extraction socket; it will be measured on the cone beam computed tomography)
Post-operative pain | 1;3;5;7;10 days
  Post-operative pain will be assessed by 10-point visual analogue scale (VAS) in the area of the extracted tooth
Post-operative oedema | 1;3;5;7;10 days
  Assessment the soft tissue epithelization using six-point Visual Analogue Scale (VAS) of swelling, where 0 indicates "no swelling", and 5 indicates "extreme severe swelling
Soft tissue epithelization | 7;10;14
  Assessment the soft tissue epithelization using a photoprotocol (the day on which full tissue regeneration has taken place will be taken into account)
Trismus | 1;3;5;7;10 days
  Assessment the distance between upper and lower incisors in mm
sRANKL (soluble receptor activator of nuclear factor-κB ligand) | before surgery, after surgery, 3;7 days
  Assessment the level of sRANKL in saliva by enzyme-linked immunosorbent assay, ELISA
OPG (osteoprotegerin) | before surgery, after surgery, 3;7 days
  Assessment the level of OPG in saliva by enzyme-linked immunosorbent assay, ELISA
Fibroblast growth factor-b (FGF-b) | before surgery, after surgery, 3;7 days
  Assessment the level of FGF-b in saliva
C-reactive protein (CRP) | before surgery, after surgery, 3;7 days
  Assessment the level of CRP in saliva by enzyme-linked immunosorbent assay
IgA | before surgery, after surgery, 3;7 days
  Assessment the level of IgA in saliva by enzyme-linked immunosorbent assay
IgG | before surgery, after surgery, 3;7 days
  Assessment the level of IgG in saliva by enzyme-linked immunosorbent assay
IgM | before surgery, after surgery, 3;7 days
  Assessment the level of IgM in saliva by enzyme-linked immunosorbent assay
Vascular endothelial growth factor (VEGF) | before surgery, after surgery, 3;7 days
  Assessment the level of VEGF in saliva by enzyme-linked immunosorbent assay

CONTACTS AND LOCATIONS:
Overall Officials: Diana Sologova, Principal Investigator — I.M. Sechenov First Moscow State Medical University (Sechenov University)

IPD SHARING:
Plan to Share IPD: No
No, dissemination of data is prohibited by the local ethics committee